CLINICAL TRIAL: NCT02424916
Title: Adoptive Transfer of CD8+ T Cells, Sorted With HLA-peptide Multimers and Specific for Melan-A and MELOE-1 Melanoma Antigens, to Metastatic Melanoma Patients. A Phase I/II, Non-randomized, Open Monocentric Study
Brief Title: Adoptive Transfer of Specific Melanoma Antigens CD8+ T Cells in Metastatic Melanoma Patients: a Phase I/II Study
Acronym: MelSort
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: UMR892 (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC12_0261
Record Dates: First submitted 2015-04-03; First posted 2015-04-23 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Melanoma
Keywords: Onco-dermatology; Adoptive transfer; Immunotherapy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous somatic cell therapy (Experimental): Patients treated with melanoma antigens-specific CD8+ T lymphocytes followed by subcutaneous injections of Proleukin.
  Interventions: Biological: Melanoma antigens-specific CD8+ T lymphocytes

INTERVENTIONS:
Biological: Melanoma antigens-specific CD8+ T lymphocytes — The intervention uses an autologous somatic cell therapy medicinal product. It consists in the intravenous injection of melanoma antigens (Melan-A and MELOE-1) - specific CD8+ T lymphocytes followed by subcutaneous injections of Proleukin.

SUMMARY:
This study evaluates the safety as well as the potential clinical efficacy of an adoptive transfer of CD8+ T cells, sorted with HLA-peptide multimers and specific for Melan-A and MELOE-1 melanoma antigens, to patients suffering from advanced metastatic melanoma (stages IIIc and IV).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 and ≤ 75 years
* Patient expressing the HLA-A*0201 subtype of the human leukocyte antigen (HLA -A2)
* Patient with metastatic melanoma stage IIIc or IV (AJCC 2010) except brain metastases
* Tumor expressing the antigens Melan-A and MELOE-1 detected by RT-PCR
* Absence of cerebral metastases
* ECOG ≤ 1 or Karnofsky ≥ 80%
* Prior adjuvant melanoma treatment (before metastatic stage) authorized (anti- BRAF, anti-CTLA4, IFN, TIL... )
* Disease measurable / evaluable within 28 days before the first administration of study treatment
* Negative viral serology (HIV 1/2, Ag p24 , HTLV 1/2 , hepatitis B and C, syphilis)
* Results of analysis:

  * Hemoglobin ≥ 10 g / dl or ≥ 6.25 mmol / l
  * Leukocytes ≥ 4000/μl
  * Lymphocytes ≥ 1500/μl
  * Platelets ≥ 80.000/μl
  * Creatinine ≤ 2.5 N
  * Total bilirubin ≤ 3 N
  * AST and ALT ≤ 3 N without liver metastases; ≤ 5 N with liver metastases
* Negative pregnancy test for women of childbearing age
* Patient affiliated to a social security system
* Patient who has signed informed consent

Exclusion Criteria:

* Brain metastases
* Ocular primitive melanoma
* Treatment of metastatic melanoma by more than two lines (chemotherapy , immunotherapy, targeted therapy or radiotherapy) or within 4 weeks before the inclusion
* Treatment with ipilimumab within 8 weeks before the inclusion
* Known allergy to albumin
* Contraindication to the use of vasopressors
* Positive viral serology for HIV 1/2 , Ag p24 , HTLV 1/2, hepatitis B or C, or syphilis
* Women who are pregnant, nursing or refusing to use contraceptives, women with no negative pregnancy test at baseline
* Presence of a second active cancer (with the exception of cervical cancer in situ or skin cancer other than melanoma)
* History of event or current event of a progressive or non-stabilized severe heart disease (congestive heart failure, coronary artery disease, uncontrolled hypertension, serious arrhythmias or ECG signs of previous myocardial infarction)
* Uncontrolled thyroid dysfunction
* Any serious acute or chronic illness (active infection requiring antibiotics, bleeding disorders or other condition requiring concomitant treatment not allowed in this study)
* History of chronic autoimmune disease (Addison's disease, multiple sclerosis, Graves' disease, rheumatoid arthritis, systemic lupus erythematosus, ... ) with the exception of patients with active vitiligo or a history of vitiligo
* History of uveitis and retinopathy associated with melanoma
* Adults under a legal protection regime (guardianship, trusteeship, "sauvegarde de justice")

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-05-26 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Clinical and biological safety defined by the NCI (Common Toxicity Criteria - Version 4.0, may 2009, http:// ctep.cancer.gov) | Until disease progression during the follow-up period of the study (12 months)
  Serious adverse effects of grade 3 and 4 will be considered to decide the suspension of inclusion

SECONDARY OUTCOMES:
Progression-free survival | From the date of the first treatment until the date of the first documented progression or the date of death from any cause, whichever came first, assessed up to 2 years
Overall survival | From the date of the first treatment until the date of death, assessed up to 2 years
Overall tumor response (complete response, partial response, stable disease) evaluated according to Response Evaluation Criteria in Solid Tumor (RECIST) and immune-related Response Criteria (irRC) | At 12 months
Duration of clinical responses defined as the time interval between the evaluation of the first objective response or stable disease and the first evaluation of disease progression | At 12 months
Persistence of injected specific T cells evaluated by immunomonitoring | At 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France